CLINICAL TRIAL: NCT02705066
Title: Citicoline Effects on Cortical Membrane Structure and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyowa Hakko Bio Co., Ltd. (Industry)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2015-8400
Record Dates: First submitted 2016-02-23; First posted 2016-03-10 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Cellulose) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo supplement
- Cognizin 250 mg/day (Experimental)
  Interventions: Dietary Supplement: Citicoline supplement
- Cognizin 500 mg/day (Experimental)
  Interventions: Dietary Supplement: Citicoline supplement

INTERVENTIONS:
Dietary Supplement: Citicoline supplement
  Other Names: Cognizin
  Arms: Cognizin 250 mg/day; Cognizin 500 mg/day
Dietary Supplement: Placebo supplement — Cellulose
  Other Names: Placebo
  Arms: Placebo (Cellulose)

SUMMARY:
The goal of this project is to determine the effects of 6-week dietary supplementation with one of two doses of citicoline (250 mg/d, 500 mg/d) or placebo on prefrontal cortical membrane dynamics (31P-MRS) and event-related functional activation (fMRI) in healthy middle-aged adults.

DETAILED DESCRIPTION:
To determine the effect of citicoline supplementation on cortical structure and function in healthy middle-aged adults. Test 1: The effect of citicoline (500 mg/d) compared with placebo on event-related anterior cingulate cortex (ACC) activation during sustained attention by fMRI. Test 2: The effect of citicoline (500 mg/d) compared with placebo on reaction time and increasing accuracy on the sustained attention task (CPT-IP). Test 3: The effect of citicoline compared with placebo on phosphodiester (PDE) and b-NTP levels in the ACC by 31P-MRS. Test 4: ACC activation and CPT-IP performance (fMRI) and ACC PDE levels (31P-MRS) following high-dose citicoline (500 mg/d) compared with placebo at Week 3. Test 5: The effect of low-dose citicoline (250 mg/d) compared with placebo on an ACC activation and CPT-IP performance (fMRI) and ACC PDE levels (31P-MRS). Test 6: Among all subjects (n=60), the relationship between baseline red blood cell (RBC) omega-3 fatty acid (EPA+DHA) levels and ACC activation, ACC PDE levels, or the effects of citicoline.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent;
* Ages 40-60 years old;
* Right handed.
* If female, not pregnant (as determined by a positive pregnancy test); and agrees to use one of the following methods of birth control: abstinence from sexual intercourse, barrier (diaphragm or condom), or oral/injectable contraceptive;

Exclusion Criteria:

* Contraindication to an MRI scan (i.e., braces, claustrophobia, pacemaker etc);
* A history of a major medical (e.g., diabetes) or neurological illness (e.g., epilepsy);
* Body mass index (BMI) ≥ 30;
* An IQ <75 and >130;
* A positive urine drug test (nicotine dependence is permitted);
* Personal history of a DSM-5 Axis I psychiatric disorder;
* Requiring treatment with a drug which might obscure the action of the study treatment.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Phosphodiester (PDE) concentrations in the ACC by 31P-MRS | 6 weeks
b-NTP concentrations in the ACC by 31P-MRS | 6 weeks

SECONDARY OUTCOMES:
Blood oxygenation level-dependent signal in the ACC during sustained attention by fMRI | 6 weeks
Reaction time (ms) on an attention task (CPT-IP) | 6 weeks
Accuracy (percent correct) on an attention task (CPT-IP) | 6 weeks

OTHER OUTCOMES:
Baseline red blood cell (RBC) omega-3 fatty acid (EPA+DHA) levels | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States